CLINICAL TRIAL: NCT01749826
Title: Inflammatory Responses to Acute and Chronic Opioid Exposure in Humans
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The cytokines in the samples were undetectable.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Larry Fu-nien Chu, Associate Professor of Anesthesia, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SU-10212009-4201
Record Dates: First submitted 2009-11-09; First posted 2012-12-17 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Inflammation
Keywords: Inflammation, opioids, immune system
MeSH Terms: conditions — Inflammation | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chronic Opioid Exposure (Experimental): 15mg sustained release morphine sulfate, with a maximum dose of 120mg. Patients will be titrated up to a maximum dose of 8 pills a day for one month.
  Interventions: Drug: Morphine Sulfate
- Acute Opioid Exposure (Experimental): 15mg sustained release morphine sulfate, with a maximum dose of 120mg. Patients will be titrated up to a maximum dose of 8 pills a day for one month.
  Interventions: Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Morphine Sulfate — 15mg sustained release morphine sulfate, with a maximum dose of 120mg. Patients will be titrated up to a maximum dose of 8 pills a day for one month.
  Other Names: MS Contin; Morphine Sulfate ER; Roxanol; Kadian

SUMMARY:
We aim to examine the extent to which inflammation is affected by acute and chronic opioid exposure.

DETAILED DESCRIPTION:
We are interested in learning how the immune system and the inflammation process is effected by acute and chronic opioid exposure. Preliminary evidence in animal models show that acute opioid exposure leads to decreased inflammatory responses, while chronic opioid exposure causes increased inflammatory responses, as measured by local cytokine release at the site of injury. Translating these findings to humans will lead to important new mechanistic knowledge that may ultimately improve our ability to treat pain.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* Healthy volunteer
* Not allergic to remifentanil

Exclusion Criteria:

* Patients younger than 18 or older than 70
* Patients unwilling or unable to follow study instructions
* Patients who don't speak English
* Patients who are taking prescription opioid medications (e.g. vicodin, percocet) or are unwilling to refrain from taking anti-inflammatory medications such as Advil or Naproxen during 2 weeks prior to and during the 1 month study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Larry Fu-nien Chu, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronic Opioid Exposure | Acute Opioid Exposure
Started | 20 | 0
Completed | 0 | 0
Not Completed | 20 | 0
Not completed — Study Terminated | 20 | 0

BASELINE CHARACTERISTICS:
Population: We were unable to perform analysis as we were unable to detect any cytokines in our samples.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Opioid Exposure | Acute Opioid Exposure | Total
Number analyzed (Participants) | 20 | 0 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (11.47) |  | 40.9 (11.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 |  | 7
  Male | 13 |  | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 3 |  | 3
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 3 |  | 3
  White | 14 |  | 14
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 |  | 20

OUTCOME MEASURES:

1. Primary Outcome: Changes in Cytokine Release
Description: 5 CCs of blood are drawn on day 1 and day 30.
Time Frame: Changes in cytokine release are compared between blood samples drawn on Day 1 and Day 30
Population: Data can not be summarized or included in this table as no data on this measure was collected. 5 CCs of blood were not drawn from any participants at any point in time during the study as the study was terminated due to a lack of resources prior to collection of any study measure data.
Arm/Group | Chronic Opioid Exposure | Acute Opioid Exposure
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Laser Doppler Images
Description: The laser doppler is a noninvasive, painless measurement of superficial perfusion that reflects inflammation. Laser doppler images will be taken once per study visit.
Time Frame: Changes in laser doppler images are measured between images taken on Day 1 and Day 30
Population: Data can not be summarized or included in this table as no data on this measure was collected. Laser doppler image data was not collected from any participants at any point in time during the study as the study was terminated due to a lack of resources prior to collection of any study measure data.
Arm/Group | Chronic Opioid Exposure | Acute Opioid Exposure
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Peltier Device-Heat Pain
Description: A hand-held 0.6x0.6 inch metal probe will be brought into contact with the patient's skin. Starting at 95 F, the probe temperature will increase at a rate of 1.8 F per second. The patient will be asked to push a button of a hand-held device as soon as the patient feels pain.
Time Frame: Differences in heat pain are assessed between measurements taken on Day 1 and Day 30
Population: Data can not be summarized or included in this table as no data on this measure was collected. Peltier device-heat pain data was not collected from any participants at any point in time during the study as the study was terminated due to a lack of resources prior to collection of any study measure data.
Arm/Group | Chronic Opioid Exposure | Acute Opioid Exposure
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mechanical Pain Stimuli
Description: Pain sensitivity will be tested with three different mechanical stimuli that can elicit mild pain:
  * Stroking stimulus: skin will be tested with a brush that is moved three times across the lesion
  * Punctuated stimulus: a metal rod (1/100 of an inch in diameter) mounted onto 10 different weights (0.03-2.9 ounces) will repetitively be placed onto the skin
  * Blunt stimulus: a flat probe (0.4 inch in diameter) will be placed five times onto the patient's skin
Time Frame: Changes in mechanical pain stimuli will be assessed between measurements taken on Day 1 and Day 30
Population: Data can not be summarized or included in this table as no data on this measure was collected. Mechanical pain stimuli data was not collected from any participants at any point in time during the study as the study was terminated due to a lack of resources prior to collection of any study measure data.
Arm/Group | Chronic Opioid Exposure | Acute Opioid Exposure
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: As no data was collected for study measures, no adverse events data was collected.
Description: There is no difference in definition. As no data was collected for study measures, no adverse events data was collected.
Arm/Group | Chronic Opioid Exposure | Acute Opioid Exposure
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
We were unable to analyze any data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No